CLINICAL TRIAL: NCT07125547
Title: Neoadjuvant Tislelizumab Combined With Nab-Paclitaxel Followed by Distal Ureterectomy for Ureteral Cancer: An Open-Label, Single-Center, Single-Arm, Phase II Clinical Trial (TRUCE-U01)
Brief Title: Neoadjuvant Tislelizumab + Nab-Paclitaxel Followed by Distal Ureterectomy for Ureteral Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRUCE-U01
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-04

CONDITIONS: Ureteral Cancer; Neoadjuvant Therapy; PD-1 Inhibitor; Kidney-sparing; Tislelizumab; Nab-paclitaxel
MeSH Terms: conditions — Ureteral Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Nab-Paclitaxel 125mg/m^2 IV on day 1 in combination with Tislelizumab 200mg IV on day 1 every 3 weeks for 2-3 cycles and then followed by distal ureterectomy (Distal ureterectomy + Partial cystectomy +Psoas hitch procedure + Ureteral reimplantation into the bladder + Ipsilateral pelvic lymph node dissection).
  Interventions: Drug: PD-1 inhibitior; Drug: Nab-paclitaxel; Procedure: distal ureterectomy

INTERVENTIONS:
Drug: PD-1 inhibitior — Tislelizumab 200mg iv will be administered on Day 1 every 3 weeks for 2-3 cycles.
Drug: Nab-paclitaxel — Nab-Paclitaxel 125mg/m2 IV will be administered on Day 1 every 3 weeks for 2-3 cycles
Procedure: distal ureterectomy — Distal ureterectomy (Distal ureterectomy + Partial cystectomy +Psoas hitch procedure + Ureteral reimplantation into the bladder + Ipsilateral pelvic lymph node dissection) will be conducted after neoadjuvant treatment.

SUMMARY:
This study is designed as an open-label, single-arm, single-center, phase II clinical trial, aiming to evaluate the efficacy and safety of neoadjuvant Tislelizumab combined with Nab-Paclitaxel followed by distal ureterectomy for patients with non-metastatic ureteral cancer (UTC). Patients enrolled will receive 2-3 cycles of Tislelizumab in combination with Nab-Paclitaxel every 3 weeks and then undergo distal ureterectomy (DU). The assessment of efficacy is based on the histology of specimen from DU, and treatment-related adverse events (TRAEs) will be recorded and evaluated according to CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged no less than 18 years old;
2. Ureteral cancer indicated by ureteroscopic biopsy and imageological examination (including CT, MRI, or PET-CT), without evidences of metastasis in chest CT scan and abdominal CT scan (T1-4N0-2M0).
3. Histologically confirmed urothelial carcinoma or urothelial carcinoma as the major pathological component >50% in the specimen from ureteroscopic biopsy;
4. Suitable and planned to receive distal ureterectomy (including distal ureterectomy + partial cystectomy + ipsilateral pelvic lymph node dissection + psoas hitch procedure + ureteral reimplantation into the bladder).
5. Expected survival time of more than 12 weeks;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2;

6.Agree to provide blood, urine, and tissue samples (for testing PD-L1 expression, tumor mutation burden, etc.); 7.The organ function levels must meet the following requirements: Hematological indicators: Absolute neutrophil count ≥1.5×10^9/L, platelet count ≥80×10^9/L, hemoglobin ≥6.0 g/dL (can be maintained through symptomatic treatment); Liver function: Total bilirubin ≤1.5 times the upper limit of normal, alanine transaminase and aspartate transaminase ≤2.5 times the upper limit of normal; Renal function: Baseline ECT renography indicates a total renal glomerular filtration rate (GFR) ≥15 ml/min, with the affected-side GFR >10 ml/min, excluding the presence of a non-functional kidney (low-level decreasing curve on dynamic renal ECT imaging) on the affected side.

8.Participants are willing to join the study and be able to sign and comply the protocol.

Exclusion Criteria:

1. Concurrent primary malignancies in other sites are excluded, except for those with a history of other malignancies that have been treated and are currently stable.
2. Confirmed bilateral upper tract urothelial carcinoma (UTUC).
3. Presence of urothelial carcinoma in the renal pelvis or bladder is excluded, except for non-muscle-invasive bladder cancer that can be completely resected via transurethral resection of bladder tumor (TURBT).
4. Received a live attenuated vaccine within 4 weeks before treatment or plan to receive during the study period;
5. Active, known or suspected history of autoimmune disease;
6. Known history of primary immunodeficiency;
7. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
8. Pregnant or breastfeeding female patients;
9. Untreated acute or chronic active Hepatitis B or Hepatitis C infection. Patients receiving antiviral therapy may be eligible if viral load is under monitored, at the discretion of the physician based on the patient's individual condition;
10. Receiving immunosuppressive medication within 4 weeks prior to starting treatment, except nasal, inhaled, topical steroids, or systemic corticosteroids at physiological doses (i.e., not exceeding 10 mg/day of prednisone or equivalent dose of other corticosteroids);
11. Known or suspected allergy to Tislelizumab or Nab-Paclitaxel;
12. Active tuberculosis;
13. Previous treatment with PD-1/PD-L1/CTLA-4 immune checkpoint inhibitors or other immunotherapies;
14. Participation in another clinical study;
15. Fertile men or women without effective contraception;
16. Uncontrolled concurrent illness, including but not limited to:

(1)HIV infection (HIV antibodies positive); (2)Uncontrolled severe infection; (3)Uncontrolled systemic disease (such as severe psychiatric, neurological disorders, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver, or kidney disease, uncontrolled hypertension [i.e., hypertension of CTCAE grade 2 or higher despite treatment]); (4)Active hemorrhage or newly developed thrombotic disease. (5)Renal failure with CKD grade 5 and undergoing dialysis treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | At the time of distal ureterectomy completed (within 14 weeks of the treatment initiated)
  Defined as no residual tumor in the specimen from distal ureterectomy.

SECONDARY OUTCOMES:
Treatment-related adverse events (TRAEs) | From neoadjuvant treatment initiation to 90 days after the last cycle of treatment.
  Treatment-related adverse events (TRAEs) ,defined as adverse events occurring from the start of treatment (C1D1) to 90 days after the completion of the last dose, including type, incidence rate, and severity grading (assessed according to the NCI-CTCAE V5.0 criteria)
Pathological Downstaging (pDS) | At the time of distal ureterectomy completed (within 14 weeks of the treatment initiated)
  Defined as a reduction in the pathological T stage and N stage of the distal ureterectomy specimen compared to the clinical T stage and N stage assessed at baseline
Objective Response (OR) | After completion of neoadjuvant therapy and before distal ureterotomy.
  Defined as the achievement of partial response (PR) or complete response (CR) based on RECIST 1.1 criteria, as assessed by imaging studies after neoadjuvant therapy.
Events-Free Survival (EFS) | up to 5 years
  Defined as the time from treatment initiated to the first occurrence of delayed surgical disease progression, local tumor recurrence (including recurrence in the upper urinary tract and bladder, excluding non-muscle-invasive bladder cancer that can be resected by TURBT), distant metastasis, or death from any cause. The study will record the 1-, 2-, and 5-year EFS rates for the target population. Kaplan-Meier methods will be used to estimate the median EFS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on EFS.
Overall Survival (OS) | up to 5 years
  Defined as the time from treatment initiated to death from any cause. The study will record the 1-, 2-, and 5-year OS rates for the target population. Kaplan-Meier methods will be used to estimate the median OS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on survival
Recurrence-Free Survival (RFS) | up to 5 years
  Defined as the time from treatment initiated to the first occurrence of tumor recurrence (including recurrence in the upper urinary tract and bladder, excluding non-muscle-invasive bladder cancer that can be removed by TURBT). The study will record the 1-, 2-, and 5-year RFS rates for the target population. Kaplan-Meier methods will be used to estimate the median RFS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on RFS.
Cancer-Specific Survival (CSS) | up to 5 years
  Defined as the time from enrollment to death caused by the tumor. The study will record the 1-, 2-, and 5-year CSS rates for the target population. Kaplan-Meier methods will be used to estimate the median CSS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on CSS.
Nephron-Sparing Survival (NSS) | up to 5 years
  Defined as the time from treatment initiated to the absence of surgical indications for nephrectomy due to upper urinary tract tumor progression or recurrence, as well as the absence of distant metastasis caused by the primary upper urinary tract tumor and death from any cause. The study will record the 1-, 2-, and 5-year NSS rates for the target population. Kaplan-Meier methods will be used to estimate the median NSS and 95% confidence interval limits, and Kaplan-Meier curves will be constructed to provide descriptive information on NSS.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tianjin Medical University, Tianjin, Outside U.S., China